CLINICAL TRIAL: NCT04749394
Title: A Phase II, Open-Label, Multi-Centre Study of Camrelizumab Plus Apatinib As Consolidation Therapy in Patients With Locally Advanced, Unresectable NSCLC, Who Have Not Progressed Following Definitive, Platinum-Based Chemoradiation Therapy
Brief Title: A Study of Camrelizumab Plus Apatinib as Consolidation Therapy in Non-Small Cell Lung Cancer Patients Treated With Chemoradiotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhouguang Hui, M.D., Chief physician, Director of VIP Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC004692
Record Dates: First submitted 2021-02-05; First posted 2021-02-11 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Locally Advanced Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Programmed cell death 1 (PD-1, PD1); Anti VEGF; Chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Camrelizumab plus apatinib as consolidation therapy
  Interventions: Drug: Camrelizumab, PD-1 monoclonal antibody; Drug: Apatinib, VEGFR2 antibody

INTERVENTIONS:
Drug: Camrelizumab, PD-1 monoclonal antibody — Camrelizumab 200mg IV, Q3W, until clinical progression/deterioration or confirmed radiological progression, or up to 1 year.
  Other Names: SHR-1210
Drug: Apatinib, VEGFR2 antibody — Apatinib 250mg PO, QD, until clinical progression/deterioration or confirmed radiological progression, or up to 1 year.
  Other Names: Apatinib Mesylate

SUMMARY:
This is a phase II, open-Label, multi-centre study to determine the efficacy and safety of Camrelizumab plus apatinib in participants with unresectable Stage III Non-Small Cell Lung Cancer (NSCLC), who have not progressed following platinum-based concurrent chemoradiation therapy (cCRT) or sequential chemoradiation therapy (sCRT). This study will be conducted in China mainland.

DETAILED DESCRIPTION:
This trial will evaluate the efficacy and safety of camrelizumab plus apatinib in participants with unresectable stage III NSCLC who have not progressed following definitive, platinum-based cCRT or sCRT. The primary endpoint is progression free survival (PFS) in the intent-to-treat (ITT) population. The secondary endpoints are as follows: 1) Overall survival (OS); 2) 1, 2, 3-year OS rates; 3) PFS rates at 12-monthand 18-month; 4) Objective response rate (ORR), 5) Duration of response (DoR); 6) Time to death or distant metastasis (TTDM); 7) Adverse effects (AEs) and severe adverse effects (SAEs) ;8) Quality of life (QoL).Exploratory objective is to explore potential biomarkers associated with efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years, male and female are not limited;
2. Patients with ECOG score of 0-1;
3. Life expectancy ≥12 weeks;
4. Patients must have histologically or cytologicallyproved NSCLC, and present with locally advanced, unresectable Stage III disease(according to 8th AJCC/UICC Classification);
5. Receipt of concurrent or sequential chemoradiation therapy which must have been completed within 42 days prior to first dose administration of the study; Consolidation chemotherapy is not permitted.
6. No progression following definitive, platinum-based, concurrent or sequential chemoradiation therapy;
7. Subject with prior anti-cancer treatment can only be enrolled when all toxicities of prior anti-cancer treatment has recovered to baseline or ≤ Grade 1, except for hearing loss, alopecia and fatigue. (according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] V5.0);
8. No prior exposure to any anti-CTLA-4, anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-VEGF treatments, as well as therapeutic anticancer vaccines;
9. Agreement to provide tumor histological specimens required for this study;
10. Adequate organ and marrow function required;
11. Fertile female were required to have a negative serum or urine pregnancy test within 72 days before the start dose of study medication; If female of childbearing potential, is willing to use adequate contraception for the course of the study through 90 days after the last dose of study medication; if male with a female partner(s) of child-bearing potential, he must agree to use adequate contraception starting with the first dose of study medication through 90 days after the last dose of study medication or have been surgically sterilized;
12. Provision of signed ICF.

Exclusion Criteria:

1. Mixed small cell lung cancer histology;
2. Disease progression after concurrent/sequential chemoradiotherapy;
3. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of treatment;
4. Receipt of live attenuated vaccine within 28 days prior to the first dose of treatment;
5. Previous enrolment of another study and receiving any study drug within 28 days prior to the first dose of treatment;
6. Patients with ≥Grade 2 pneumonitis from the prior anti-cancerchemoradiation therapy;
7. Imaging (CT or MRI) shows the tumor invading large vessels or blurring the boundary with vessels;
8. History of organ transplant or allogeneic hematopoietic stem cell transplantation;
9. Patients with any active autoimmune disease or history of autoimmune disease;
10. Patients with innate or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection;
11. Uuntreated active hepatitis B or, hepatitis C or active tuberculosis or currently receiving anti-tuberculosis treatment co-infection with hepatitis B and hepatitis C;
12. Subjects receiving systemic treatment with corticosteroids (>10mg/day of prednisone or its equivalent) or other immunosuppressants within 14 days prior to the first administration;
13. History of another primary malignancy within 5 years prior to enrollment, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study;
14. Pulmonary function test: FEV1< 1.2L or DLCO < 50% of predicted value;
15. Patients with cardiac insufficiencyheart diseases including: 1) NYHA III-IV; 2）Acute coronary syndrome; 3) Supraventricular or ventricular arrhythmias requiring clinical intervention; 4) Pericardial and myocardial diseases; 5) Echocardiography indicates that the left ventricular ejection fraction (LVEF) is < 50%;
16. Patients with uncontrollable hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, despite the best drug treatment);
17. Patients who have had arteriovenous thrombosis events within 6 months, such as cerebrovascular accident (including cerebral embolism, deep vein thrombosis, pulmonary embolismcerebral hemorrhage, cerebral infarction, transient ischemic attack, etc.);
18. Patients with hemoptysis, active bleeding, ulcer, intestinal perforation and intestinal obstruction within 3 months before administration;
19. Significant hemoptysis symptoms or daily amount of hemoptysis up to 2.5mL or more within 30 days before the first administration;
20. Known hereditary or acquired bleeding and thrombosis tendency (such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.);
21. Routine urine test indicated that urine protein was ≥ (++), or 24-hour urine protein was ≥ 1g, or severe liver and kidney dysfunction;
22. Patients with severe infection or fever of unknown origin > 38.5 degrees C within 24 weeks before medication;
23. Pregnant or lactating women; those with fertility who are unwilling or unable to take effective contraceptive measures;
24. Known allergies, hypersensitivity, or intolerance to camrelizumab or its excipients, apatinib and chemotherapy drugs;
25. Any conditions, judged by investigators, that may impair the subject or cause the subject to be unable to meet or perform the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | From the first date of treatment until the date of objective disease progression or death (up to maximum 24 months)
  PFS is determined by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Overall Survival (OS) | up to approximately 36 months
  OS is defined as the first date of treatment to date of death from any causes.
PFS at 12 months (PFS12) | up to maximum 12 months
  PFS will be calculated using Kaplan-Meier product limit methods.
PFS at 18 months (PFS18) | up to maximum 18 months
  PFS will be calculated using Kaplan-Meier product limit methods.
OS at 12 months (OS12) | up to maximum 12 months
  OS will be calculated using Kaplan-Meier product limit methods.
OS at 24 months (OS24) | up to maximum 24 months
  OS will be calculated using Kaplan-Meier product limit methods.
OS at 36 months (OS36) | up to maximum 36 months
  OS will be calculated using Kaplan-Meier product limit methods.
Objective response rate (ORR) | up to approximately 24 months
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 by investigator.
Duration of Response (DoR) | up to approximately 24 months
  DoR is defined as the first date of treatment to the progression, or the last evaluable assessment in the absence of progression.
TTDM | up to approximately 36 months
  TTDM is defined as the first date of treatment to the first date of distant metastasis or death in the absence of distant metastasis.
Number of participants with AEs, SAEs, Treatment-related Adverse Events (TRAEs). | From screening (Day -28) till final visit (up to a maximum of 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No